CLINICAL TRIAL: NCT06627270
Title: A Phase II Single-arm Cohort Study Establishing the Effect of Antibiotic Treatment on Intratumoral Bacteria in Surgical Patients With Oral Cancer
Brief Title: Antibiotic Treatment Effects on Intratumoral Bacteria Modulation in Surgical Patients With Oral Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6324
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Oral Squamous Cell Carcinoma; Oral Cancer; Head and Neck Cancer; Head and Neck Carcinoma
Keywords: Metronidazole; Chlorhexidine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Head and Neck Neoplasms | interventions — Metronidazole; Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 days of metronidazole and chlorhexidine (Experimental): Participants will receive metronidazole (500 mg t.i.d. x 10 days) and chlorhexidine (10 ml t.i.d. x 10 days) prior to surgical resection.
  Interventions: Drug: Metronidazole; Other: Chlorhexidine

INTERVENTIONS:
Drug: Metronidazole — Participants will receive metronidazole (500 mg t.i.d. x 10 days)
Other: Chlorhexidine — Mouth rinse chlorhexidine (10 ml t.i.d. x 10 days)
  Other Names: CHX

SUMMARY:
The goal of this phase II single arm clinical study is to evaluate the effect of antibiotics (metronidazole) and oral chlorhexidine (CHX) in reducing the bacteria load within tumors of patients undergoing surgery for oral cancer.

DETAILED DESCRIPTION:
The prognosis for patients with locally advanced, non-Human Papillomavirus (HPV) associated head and neck squamous cell carcinoma (HNSCC) remains poor. The immunosuppressive tumor immune microenvironment in HNSCC presents a significant barrier to both conventional and immune-based therapies. Recent studies have indicated that dysbiotic oral microbiota, particularly in the context of periodontal disease, can contribute to chronic oral mucosal inflammation and the recruitment of suppressive immune cell infiltrates. Bacterial-induced chronic inflammation may play a crucial role in treatment resistance in HNSCC. Understanding the impact of microbial modulation on the tumor immune microenvironment in HNSCC could lead to the identification of novel therapeutic targets.

In this single-arm phase II clinical trial, oral cancer patients will be treated with oral metronidazole and CHX rinses prior to surgery. Investigator will assess the ability for the treatment to reduce the absolute amount of intratumoral bacteria and evaluate changes in the intratumoral bacterial community and infiltrating immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed squamous cell carcinoma of the oral cavity
* Must have planned surgery for curative intent
* Participants ≥ 18 years of age
* Participants must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Known allergy to metronidazole and/or chlorhexidine
* Severe liver or kidney disease as determined by history of laboratory tests
* Participants actively drinking alcohol (unable to abstain for the 10 day antibiotic period)
* Recurrent oral cancer after prior radiation or chemoradiation
* Participants with unresectable oral cancer
* Participants unable to tolerate and/or absorb oral medication
* Participants currently or have taken other antibiotics within the prior 60 days
* Participant is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in absolute amount of intraumoral bacteria as quantified by 16S rRNA qPCR | Baseline, surgery (10 days post intervention)
  The difference between pre-treatment and post-treatment tumor bacteria burden will be assessed.

SECONDARY OUTCOMES:
Change in absolute amount of intraumoral bacteria in post treatment participants compared to control patients as quantified by 16S rRNA qPCR | Baseline, surgery (10 days post intervention)
Disease-free survival | Time from date of randomization to recurrence, second primary malignancy, or death, as determined by standard of care surveillance, up to three years.
Overall Survival | Time from date of randomization to recurrence, second primary malignancy, or death, as determined by standard of care surveillance, up to three years.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Silver, MD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic Foundation
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
RNAseq results will be shared upon publication, not patient identifiers will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the time of publication or after 3 years